CLINICAL TRIAL: NCT01494571
Title: Pediatric Optimization of the PharmaJet Needle-Free Intradermal Delivery System
Acronym: PharmaJet
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1362
Record Dates: First submitted 2011-12-12; First posted 2011-12-19 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2012-12

CONDITIONS: Functionality and Performance of Device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- 90 pediatric, 7 to 14 year old subjects
- 30 pediatric, 5 to 6 year old subjects
- 30 pediatric, 3 to 4 year old subjects
- 30 pediatric, 1 to 2 year old subjects
- 30 pediatric, 6 to 12 month old subjects
- 30 pediatric, 4 to 6 month old subjects
- 30 pediatric, 2 to 4 month old subjects

SUMMARY:
The PharmaJet needle-free injection system is a consistent approach to delivering injectates into the dermal layer of the human skin for the purpose of vaccination or medication delivery.

DETAILED DESCRIPTION:
Up to 400 children, ages 2 months through 14 years

1. To assess measures of injection performance, including estimates of injection completeness by collecting residual surface moisture with filter paper that will be circled with indelible ink; the volume will be compared to a reference set of moisture recordings.
2. To document completeness of injections; completeness is defined as <10% of 0.1 ml volume remaining on the skin surface immediately after injection. Measurement of the bleb size following injection will recorded in millimeters.
3. To ensure device is well received by subjects. Subject's response to the injection will be noted by the subject and/or family members after the procedure for up to 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children between ages 2 months and 14 years
* Outpatient, expected to go home day of surgery
* Written consent and assent when appropriate
* Willing to complete and return pain diary (postcard) after 48 hours

Exclusion Criteria:

* Presently have skin rash at the intended injection site
* Have a history of use of any topical or systemic medications at the intended injection site that could have potentially altered the normal physical properties of the skin (i.e. atrophy from chronic steroid use, thinning of the skin from topical or systemic retinoids).
* Have a permanent physical change in the skin at the intended injection site, such as burns, scars or prior radiation therapy.
* Skin disorders that may predispose them to develop skin lesions at sites of trauma.
* Present use of any blood thinning medications.
* In the 10-11 year old cohort, none of the participants can have started puberty.

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 400 children, aged 2 months to 14 years
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Completeness of injection | within one minute after injection
  To assess measures of injection performance, including estimates of injection completeness by collecting residual surface moisture with filter paper that will be circled with indelible ink; the volume will be compared to a reference set of moisture recordings. Measurement of the bleb size following injection will recorded in millimeters.
Size of bleb on skin after injection | within 2 minutes after injection
  Measurement of the bleb size immediately following injection will be determined using a millimeter ruler
Acceptability by subject | up to 48 hrs
  subjects response to the injection-level of pain or discomfort. Subjects response will not be collected for those who opt to receive the injections while under anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Galinkin, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States